CLINICAL TRIAL: NCT06818188
Title: Effect of Rhythmic Auditory Stimulation(RAS) on Turning in Post-stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/62
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: post stroke; rhythmic auditory stimulation; turning based specific training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Turning based training without RAS (Active Comparator): The participants will receive turning based training without RAS, 3 days per week on alternate days for turning, balance and gait improvement.
  Interventions: Other: Turning based specific training without rhythmic auditory stimulation (RAS)
- Turning based training with RAS (Experimental): The participants will receive turning based training with RAS, 3 days per week on alternate days for turning, balance and gait improvement.
  Interventions: Other: Turning based specific training with rhythmic auditory stimulation (RAS)

INTERVENTIONS:
Other: Turning based specific training with rhythmic auditory stimulation (RAS) — The study involved an experimental group that underwent a 6-week turning-based training with rhythmic auditory stimulation (TBST-RAS), performed three times a week on alternate days. The purpose was to improve motor control and walking abilities through rhythmic auditory cues, specifically adjusting the metronome's beat to the patient's cadence.
  Week 1: Patients performed turning exercises around a cone and walking with visual cues at 5% rhythmic auditory cue intensity, with rest periods.
  Weeks 2-3: The intensity of rhythmic auditory cues increased to 10%, and patients engaged in cone turning, figure-of-eight walking, and walking with visual cues, with rest breaks in between.
  Weeks 4-5: Rhythmic auditory cue intensity increased to 15%. Exercises included cone turning, figure-of-eight walking, walking with visual cues, multidirectional stepping, and rest periods.
  Week 6: The final week involved exercises with a further increase in rhythmic auditory cue intensity to 20%. The exercise
  Arms: Turning based training with RAS
Other: Turning based specific training without rhythmic auditory stimulation (RAS) — The control group underwent 6 weeks of turning-based specific training without rhythmic auditory stimulation (TBST), performed three times a week on alternate days. The training followed this pattern:
  Week 1: Patients began with cone turning for 5 minutes, followed by 2 minutes of rest. Then, they walked with visual cues for 5 minutes, also without rhythmic auditory stimulation.
  Weeks 2-3: The exercises continued with cone turning and figure-of-eight walking for 5 minutes each, with 2-minute rest periods in between. Patients also walked with visual cues for 5 minutes without RAS.
  Weeks 4-5: The exercises included cone turning, figure-of-eight walking, walking with visual cues, and multidirectional stepping (forward, backward, laterally), all for 5 minutes each, with rest periods between exercises.
  Week 6: In the final week, the duration of cone turning and figure-of-eight walking was reduced to 3 minutes, but the exercises still had 2-minute rest periods in between. Patients also p
  Arms: Turning based training without RAS

SUMMARY:
As, stroke is the second leading cause of death and disability globally, leads to postural changes, disturbance in balance, increase fall risks, & gait dysfunctions, affecting daily activities and walking ability.As, turning is the major component of ambulation. But this difficulty in post stroke results in increased fall risk.Stroke survivors encounter multiple gait abnormalities, which increases difficulty in changing direction.Multiple studies have reported that, RAS with beats of metronome is an effective intervention on balance & gait patterns i-e stride length, gait speed, & symmetry in post-stroke patients .With little evidence available targeting comparative effectiveness with & without RAS on turning in post-stroke patients. This study will fill this gap, to determine the effect on changing direction, with & without RAS and will be helpful in providing evidence to literature, will provide treatment protocol for turning in gait.

DETAILED DESCRIPTION:
CHAPTER III OBJECTIVES OF STUDY

1. To determine the effect on turning in post-stroke patients with and without rhythmic auditory stimulation (RAS)
2. To determine the effect on balance in post-stroke patients with and without rhythmic auditory stimulation (RAS)
3. To determine the effect on cadence in post-stroke patients with and without rhythmic auditory stimulation (RAS)
4. To determine the effect on gait speed in post-stroke patients with and without rhythmic auditory stimulation (RAS)

HYPOTHESIS OF STUDY

ALTERNATE HYPOTHESIS:

1. HA: There is a statistically significant difference on turning in post-stroke patients with and without RAS i-e P<0.5
2. HA: There is a statistically significant difference on balance in post-stroke patients with and without RAS i-e P<0.5
3. HA: There is a statistically significant difference on cadence in post-stroke patients with and without RAS i-e P<0.5 4:HA: There is a statistically significant difference on gait speed in post-stroke patients with and without RAS i-e P<0.5

NULL HYPOTHESIS:

1. HO: There is no statistically significant difference on turning in post-stroke patients with and without RAS i-e P>0.5
2. HO: There is no statistically significant difference on balance in post-stroke patients with and without RAS i-e P>0.5
3. HO: There is no statistically significant difference on cadence in post-stroke patients with and without RAS i-e P>0.5
4. HO: There is no statistically significant difference on gait speed in post-stroke patients with and without RAS i-e P>0.5

Sample Selection Criteria:

Recruitment was based on the inclusion and exclusion criteria, as below:

Inclusion Criteria:

Age 45-60 years Male and Females both Sub-acute and chronic ischemic stroke patient (MCA >6months) Mini Mental State Examination score of 25 or higher Functional Ambulation Category (2-3) Berg Balance scale, score of 40-50

Exclusion Criteria:

Hemorrhagic stroke Case or history of epilepsy Patients, having other neurological conditions, Alzheimer, Parkinson & Dementias

RANDOMIZATION & ALLOCATION:

Recruited participants were allocated to the experimental and the control group through simple random sampling technique using coin toss method.

Experimental group has received Turning based specific training with Rhythmic Auditory Stimulation (TBST-RAS).

Control group has received Turning based specific training without Rhythmic Auditory Stimulation (TBST).

BLINDING:

This study was non-blinded.

DATA COLLECTION PROCEDURE:

Before commencing data collection, we obtained ethical approval from ERC Foundation University Islamabad, following which approval from the higher authorities of Fauji Foundation Hospital Rawalpindi was taken. Participants were approached during their free time and referred by medical OPD who were willing to volunteer for the study. Informed consent in written form was taken after explaining the research purpose along with the associated participation benefits and risks to the individuals. Participants were included in the study after considering inclusion and exclusion criteria. Baseline data was obtained, by performing 180 degree test, Figure of eight, Berg balance scale, Time up and Go (TUG), and 10 meter walk (10MWT) for Turning, Balance, Cadence, and Gait Speed respectively, then participants underwent an intervention phase of 6 weeks (3 days per week on alternate days). After completion of sessions, post-assessment was done for evaluation of turning, balance and gait.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-60 years
* Male & Females both
* Sub-acute & chronic ischemic stroke patient (MCA >6months)
* Mini Mental State Examination score of 25 or higher
* Functional Ambulation Category score 2-3
* Berg Balance scale score of 40-50

Exclusion Criteria:

* Hemorrhagic stroke
* Case or history of epilepsy
* Patients, having other neurological conditions, Alzheimer, Parkinson & Dementias

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Turning assessment | 6 weeks
  180 degree turn test will be used. piece of colored tape placed on floor to mark starting point, participant will be asked to turn 180° on spot from standing start position & within a designated marked area on floor.
  The starting point is marked with a piece of colorful tape on the floor, and the participant is then told to stand with their feet pointed in that direction. After that, they are then instructed to immediately turn 180 degrees from the starting position while standing in a certain, indicated area on the floor. The number of steps required to turn 180 degrees will be counted after the subject is instructed to turn "as fast as he/she can." There will be three rotations in each direction, with a one-minute of break in between. The chance of falling increases with more than five steps. About three seconds is the meantime
Turning assessment | 6 weeks
  Through figure of 8. participant will walk in figure of 8 shape around 2 cones (Clockwise & anti-clockwise)
Balance | 6 weeks
  The Berg Balance Scale is 14 item scale, assesses the balance of patients with neurological disorders. Performance is assessed on different tasks and each task is graded with a 5- point ordinal scale ranging from 0 to 4, Maximum score à 56 points à adequate postural balance & no risk of falls. Score equal to or less than 45 points indicates risk of fall. Between 56 & 41 points, indicate a low risk of falling, between 40 & 21 points a medium risk of falling, & between 20 and 0 points a high risk of falling.
Balance | 6 weeks
  Timed up and go test. It measures the time taken for an individual to rise from a chair, walk 3 meters, turn, walk back and sit down
Cadence | 6 weeks
  10 meter walk test
Gait speed | 6 weeks
  10 meter walk test. Mark off 10 m on floor with tape, time in sec how long it takes for patient to walk in 10 meter, having them start few feet before the line and keep going a few feet after the line. calculate in Meters/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan